CLINICAL TRIAL: NCT04839016
Title: A Randomized, Double-blind, Multicenter, Placebo-controlled, Phase III Adaptive Study of SHR-1314 to Assess Efficacy and Safety in Patients With Moderate-to-Severe Plaque Psoriasis
Brief Title: Efficacy 、Safety and PK of SHR-1314 in Patients With Moderate-to-Severe Plaque Psoriasis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHR-1314-301
Record Dates: First submitted 2021-04-08; First posted 2021-04-09 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Moderate-to-Severe Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment group A (Experimental)
  Interventions: Drug: SHR-1314
- Treatment group B (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SHR-1314 — SHR-1314
  Arms: Treatment group A
Drug: Placebo — Placebo
  Arms: Treatment group B

SUMMARY:
The purpose of this study is to assess efficacy, safety, pharmacokinetics and immunogenicity of subcutaneous SHR-1314 in Patients with Moderate-to-Severe Plaque Psoriasis

ELIGIBILITY:
Inclusion Criteria:

1. Men or women at least 18 years of age at time of screening.
2. Chronic plaque-type psoriasis present for at least 6 months and diagnosed before randomization.
3. Moderate to severe psoriasis as defined at Baseline/ randomization by:

   PASI score of 12 or greater, and sPGA score of 3 or greater (based on a static scale of 0 - 5), and Body Surface Area (BSA) affected by plaque psoriasis of 10% or greater.
4. Subject has moderate to severe chronic plaque-type psoriasis that is inadequately controlled by topical treatment and/or phototherapy and/or previous systemic therapy.
5. Body Mass Index (BMI) is 18 kg/m2 or above at screening

Exclusion Criteria:

1. Forms of psoriasis other than chronic plaque-type (e.g., pustular, erythrodermic and guttate psoriasis) at Screening or Baseline/randomization.
2. Drug-induced psoriasis.
3. Had a clinically significant flare of psoriasis during the 12 weeks prior to baseline (Week 0).
4. Presence of other skin conditions (e.g. skin infections, seborrheic dermatitis) that in the judgement of the Investigator could interfere with assessment of psoriasis.
5. History of inflammatory bowel disease or have other ongoing active autoimmune diseases.
6. At screening, history or symptoms of malignancy of any organ system, treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
7. History of congestive heart failure (New York Heart Association [NYHA] functional classification ≥III), cerebro-cardiovascular events, or serious bleeding events at screening and / or randomization that in the judgement of the Investigator prevents the subject from participating in the study.
8. Active systemic infections (other than common cold) during the 4 weeks before randomization (e.g., hepatitis), or serious infections requiring hospitalization and/or intravenous injection of antibiotic treatment within eight weeks prior torandomization.
9. History of depression and/or suicidal ideation or any suicidal behavior based on an assessment with the Columbina Suicide Severity Rating Scale (C-SSRS) at screening and baseline (Posner K et al, 2011), The subjects will be exluded if any answer to question is "yes" in the questionnaire orare clinically judged by the investigator to be at risk for suicide.
10. All subjects will be tested for tuberculosis status using IGRA and X-ray test.
11. Have evidence of positive test for hepatitis B, hepatitis C antibody, or human immunodeficiency virus (HIV) antibodies.
12. Have a known allergy or hypersensitivity to any biologic therapy at screening that would pose an unacceptable risk to the subject if participating in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 660 (Estimated)
Dates: Start 2021-04-25 (Estimated); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects who achieve at least 90% improvement in PASI score (PASI 90) at Week 12 | Week 12
sPGA of 0 or 1 response at Week 12 | Week 12

SECONDARY OUTCOMES:
Percentage of subjects who achieve at least 75% improvement in PASI score (PASI 75) at Week 12； | Week 12；
Percentage of subjects who achieve at least 100% improvement in PASI score (PASI 100) at Week 12 | Week 12
sPGA of 0 response at Week 12 | Week 12